CLINICAL TRIAL: NCT03537846
Title: Osteoporosis Awareness Survey of Women in Champagne Ardenne
Acronym: MPCosteoporose
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18048
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteoporosis and women: Patient women over thirty years old

SUMMARY:
Osteoporosis is characterized by low bone mineral density and alterations in bone microarchitecture, leading to bone fragility and high risk of fractures. In the peri-menopausal period and during menopause, estrogen deficiency is responsible for an acceleration of bone remodeling. It is therefore important to sensitize women to this pathology at the beginning of menopause.

Osteoporosis is a public health issue with more than 3 million women in France suffering from almost ¼ of the population over 50 years old. Paradoxically, the number of bone densitometry and prescribed osteoporosis drugs are decreasing. There is an under-screening and a disinterest of the pathology on the part of the medical world and the patients.

The investigators hypothesize that women lack knowledge about osteoporosis. This study will identify these gaps, and put in place appropriate strategies to improve this knowledge.

For this purpose, a descriptive cross-sectional observational study will carry out, through the fulfillment of self-administered questionnaire for women over 30 years old. The main objective is to assess the knowledge of women, about osteoporosis and its consequences. The judgment criterion is based on a percentage of correct answers per question. The interests of the study are to identify gaps in knowledge, to optimize the investigator's therapeutic education, to fight patient wait-and-see and false beliefs, and finally to improve adherence and longer-term adherence.

DETAILED DESCRIPTION:
This is a descriptive cross-sectional observational study, recruiting women over 30 years old, by the diffusion of the questionnaire in the general practices of Champagne-Ardenne, and the rheumatology department of CHU de Reims.

The main objective of the study is to assess the knowledge of women over 30 on osteoporosis and its consequences. The judgment criterion is a calculation of the percentage of correct answers per question. The investigation plan is based on a self-administered questionnaire survey .The statistical analysis plan is based on a descriptive analysis with sorting flat and sorted; The questionnaires will be disseminated from March 2018 to May 2018, with the valuation of results on June 1, 2018.

This questionnaire includes:

* 6 questions relating to the patient : risk of osteoporosis and specific management.
* 17 questions about osteoporosis knowledge
* 8 questions about information resources received on osteoporosis ( media, general practitioner …) The questionnaire will be accompanied by a cover letter and a consent form. The filling of the questionnaire should last between 5 and 7 minutes. The patient will then give back the questionnaire directly to the person who has offered him to fill it out (general practitioner, rheumatologist, nurse).

The questionnaires will be placed in waiting rooms of doctors, dentists, and paramedics of the Marne, the Ardennes, and the Aube.

ELIGIBILITY:
inclusion criteria :

* gender : women
* age over thirty years old

exclusion criteria :

* Cognitive state incompatible with the collection of information
* women doctors

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity
Study Population: women
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis with sorting flat and crossed sorting and calculation percentage | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided